CLINICAL TRIAL: NCT01450865
Title: Evaluation of the Effect of the K+-Channel Opener Flupirtine on the Excitability of Human Peripheral Myelinated Axons in Vivo: a Randomised Controlled Trial
Brief Title: Effect of the Kv7-channel Opener Flupirtine on the Excitability of Human Peripheral Myelinated Axons in Vivo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Johannes Fleckenstein, Registrar, MD, Multidisciplinary Pain Centre, Department of Anaesthesiology, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: EudraCT 2007-007314-10
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Axonal Change, Neuronal; Pain
Keywords: neuropathy; axonal excitability; myelinated nerve; human; ectopic discharge; flupirtine
MeSH Terms: conditions — Pain | interventions — flupirtine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo first (Experimental): Volunteers receive placebo first and after a cross-over period of at least 7 days flupirtine second. On the days of the experiment outcome is taken as the change in excitability from Baseline (all measures before intervention) to a timepoint two hours after intervention
  Interventions: Drug: flupirtine
- Flupirtine first (Experimental): Volunteers receive flupirtine first and after a cross-over period of at least 7 days placebo second. On the days of the experiment outcome is taken as the change in excitability from Baseline (all measures before intervention) to a timepoint two hours after intervention
  Interventions: Drug: flupirtine

INTERVENTIONS:
Drug: flupirtine — Potassium channel opener (SNEPCO)
  Other Names: brand names: Trancopal Dolo, Katadolon

SUMMARY:
Slow axonal Kv7 potassium channels are found along unmyelinated axons and at the nodes of Ranvier of myelinated axons in peripheral nerve. As such the pharmacological activation of Kv7 channels offers a potential means of reducing the excitability of peripheral axons. To determine whether this is the case for human peripheral myelinated axons, the effect of the Kv7 channel agonist flupirtine on the electrical excitability of A fibres was examined in both isolated segments of human sural nerve in vitro and in motor axons of the median nerve supplying abductor pollicus brevis in vivo. Axonal excitability was assessed in 21 human sural nerve fascicles in vitro and in 20 volunteers in vivo using threshold tracking in QTRAC (© Institute of Neurology, London, UK). Strength-duration time constant, rheobase current, relative refractory period (RRP), post spike superexcitability at 5 and 7 ms and threshold electrotonus over the 90 100 ms period were used as indices of electrical excitability. In addition, suppression of ectopic discharge in a model of upper limb ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily
* age > 18 years old

Exclusion Criteria:

* current use of medication (e.g. analgetics, antiepileptics, antidepressants, etc.)
* prevailing organic disease (e.g. diabetes, vascular or neurologic illness, etc.)
* previous physical trauma of the forearm (e.g. burning, surgery)
* primary organ failure
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Axonal Excitability as assessed with QTrac | Change of neuronal excitability from Baseline (before) to two hours after intervention
  The primary outcome parameter of axonal excitability was the relative refractory period (RRP) as assessed with threshold tracking techniques. Strength-duration time constant, rheobase current, refractoriness determined at 2 and 2.5 ms, superexcitability at 7 ms and threshold electrotonus over the 90 100 ms period were used as secondary outcome measures.

SECONDARY OUTCOMES:
Ectopic Discharge | Change of neuronal excitability from Baseline (before) to two hours after intervention
  Further secondary outcome measures were power content for the surface EMG and the ranked summed scores for the McGill pain questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Irnich, MD, PhD, Principal Investigator — Multidisciplinary Pain Unit Department of Anaesthesiology University of Munich Pettenkoferstr. 8a D-80336 Munich
Locations (1):
- Multidisciplinary Pain Unit Department of Anaesthesiology University of Munich Pettenkoferstr. 8a, Munich, Bavaria, Germany

REFERENCES:
- [Result] Fleckenstein J, Sittl R, Averbeck B, Lang PM, Irnich D, Carr RW. Activation of axonal Kv7 channels in human peripheral nerve by flupirtine but not placebo - therapeutic potential for peripheral neuropathies: results of a randomised controlled trial. J Transl Med. 2013 Feb 8;11:34. doi: 10.1186/1479-5876-11-34. PMID 23394517
- See also: Homepage of the respective Journal — http://www.translational-medicine.com/content/11/1/34